CLINICAL TRIAL: NCT03624595
Title: Effect of Low-dose Dexmedetomidine on Postoperative Delirium in Patients After Cardiac Surgery: A Multicenter, Double-blinded, Randomized Controlled Trial
Brief Title: Low-dose Dexmedetomidine and Postoperative Delirium After Cardiac Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-Xin Wang (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Sponsor-Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology and Critical Care Medicine, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-181
Record Dates: First submitted 2018-08-05; First posted 2018-08-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; Dexmedetomidine; Delirium; Survival
Keywords: Cardiac Surgery; Cardiopulmonary Bypass; Dexmedetomidine; Delirium; Survival
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine infusion is administered from 16:00 to 08:00 during the night of surgery; and will repeated for a maximum of 5 consecutive nights. For patients with mechanical ventilation, the infusion rate is 0.2-0.7 ug/kg/h; for those without mechanical ventilation, the infusion rate is 0.05-0.2 ug/kg/h. The target depth of sedation is Richmond Agitation-Sedation Scale (RASS) -1.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Placebo (normal saline) infusion is administered from 16:00 to 08:00 in the same speed for the same duration as in the dexmedetomidine group. The conventional sedation is provided when necessary with propofol and/or midazolam by intravenous infusion/injection. The target depth of sedation depth is RASS -1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion is administered from 16:00 to 08:00 during the night of surgery in the intensive care unit; and will repeated for a maximum of 5 consecutive nights. For patients with mechanical ventilation, the infusion rate is 0.2-0.7 ug/kg/h; for those without mechanical ventilation, the infusion rate is 0.05-0.2 ug/kg/h. The target depth of sedation is Richmond Agitation-Sedation Scale (RASS) -1.
  Other Names: Low-dose dexmedetomidine infusion
  Arms: Dexmedetomidine group
Drug: Placebo — Placebo (normal saline) infusion is administered in the same rate for the same duration as in the dexmedetomidine group. The conventional sedation is provided when necessary with propofol and/or midazolam by intravenous infusion/injection. The target depth of sedation depth is RASS -1.
  Other Names: Normal saline infusion
  Arms: Placebo group

SUMMARY:
Delirium is an acutely occurred and fluctuating cerebral dysfunction characterized with inattention, altered consciousness, cognitive decline and/or abnormal perception. It is common in the elderly after cardiac surgery and is associated with worse outcomes. Causes leading to delirium are multifactorial but sleep disturbances remains an important one. In previous studies, sedative-dose dexmedetomidine improves sleep quality in ICU patients with mechanical ventilation; and low-dose dexmedetomidine improves sleep quality in postoperative patients without mechanical ventilation. In recent studies of elderly after noncardiac surgery, night-time infusion of low-dose dexmedetomidine reduces delirium and improves 2-year survival. The investigators hypothesize that, for elderly patients after cardiac surgery, night-time infusion of dexmedetomidine may also improve sleep quality, reduce delirium development and improve 2-year survival.

DETAILED DESCRIPTION:
Delirium is an acutely occurred and fluctuating cerebral dysfunction characterized with inattention, altered consciousness, cognitive decline and/or abnormal perception. It is common in the elderly after cardiac surgery and is associated with worse outcomes.

The development of delirium is a consequence of multiple factors. For patients undergoing cardiac surgery, surgical stress and/or cardiopulmonary bypass can produce hyper-inflammatory and stress response, both of which are important factors leading to delirium. Meanwhile, patients in ICU after major surgery often develop sleep disturbances, which are also associated with increased risk of delirium.

Dexmedetomidine is a highly selective α2-adrenoceptor agonist with sedative, analgesic and anxiolytic properties. In previous studies of elderly patients admitted to ICU after non-cardiac surgery, continuous infusion of low-dose dexmedetomidine during nighttime improves sleep quality, reduces delirium, and improves 2-year survival.

The investigators hypothesize that, for patients admitted to ICU after cardiac surgery, nighttime infusion of low-dose dexmedetomidine can decrease the incidence of delirium and improve long-term survival. The purpose of this study is to investigate the effect of nighttime infusion of low-dose dexmedetomidine on postoperative sleep quality, delirium, and 2-year survival in elderly patients admitted to ICU after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years but <90 years;
2. Scheduled to undergo cardiac surgery with cardiopulmonary bypass under general anesthesia;
3. Expected to stay in the intensive care unit (ICU) for at least 1 night after surgery.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded.

1. Refuse to participate in the study;
2. Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
3. Preoperative obstructive sleep apnea (previously diagnosed as obstructive sleep apnea, or the snoring, tiredness, observed apnea, high blood pressure-body mass index, age, neck circumference and gender [STOP-Bang] questionnaires ≥3);
4. Inability to communicate during the preoperative period because of coma, profound dementia or language barrier;
5. Preoperative sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree atrioventricular block or above without pacemaker;
6. Severe hepatic dysfunction (Child-Pugh class C);
7. Severe renal dysfunction (requirement of renal replacement therapy) before surgery;
8. Presence of delirium (diagnosed by the Confusion Assessment Method [CAM]/CAM for the Intensive Care Unit [CAM-ICU]);
9. Current treatment with dexmedetomidine or clonidine.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium within the first 5 days after surgery | During the first 5 days after surgery
  Delirium is assessed twice daily (8:00-10:00 am, 18:00-20:00 pm) with the Confusion Assessment Method (CAM, for patients without mechanical ventilation) or CAM for the intensive care unit (CAM-ICU, for patients with mechanical ventilation) during postoperative days 1-5.

SECONDARY OUTCOMES:
Duration of mechanical ventilation after surgery | Up to 30 days after surgery
  Duration of mechanical ventilation after surgery
Length of stay in ICU after surgery | Up to 30 days after surgery
  Length of stay in ICU after surgery
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of Major Adverse Cardiovascular Events (MACEs) within 30 days after surgery | Up to 30 days after surgery
  Postoperative Major Adverse Cardiac Events (MACEs) include in-hospital death, myocardial infarction, second surgery, non-fetal cardiac arrest/ventricular fibrillation, and stroke. The occurrence of major postoperative events is followed up twice daily during postoperative days 1-5, then once a week until 30 days after surgery.
Incidence of other complications | Up to 30 days after surgery
  Incidence of other complications (including hospital re-admission) within 30 days after surgery.
All-cause 30-day mortality | At 30 days after surgery
  All-cause mortality within 30 days after surgery
Subjective sleep quality at 30 days after surgery | At 30 days after surgery
  Subjective sleep quality at 30 days after surgery is assessed with Pittsburgh sleep quality index (PSQI)
2 -year Major Adverse Cardiac and Cerebrovascular Events (MACCEs)-free survival after surgery | Up to 2 years after surgery
  Major Adverse Cardiac and Cerebrovascular Events (MACCEs) include cardiac death, myocardial infarction, revascularization, and stroke.
2-year overall survival after surgery | Up to 2 years after surgery
  2-year survival overall after surgery
Cognitive function in 1- and 2-year survivors | At the end of the 1st and 2nd years after surgery
  Cognitive function in 1- and 2-year survivors is assessed with the modified Telephone Interview for Cognitive Status (TICS-m, score ranges from 0 to 40, with higher score indicating better function).
Quality of life in 1- and 2- year survivors | At the end of the 1st and 2nd years after surgery
  Quality of life in 1- and 2-year survivors is assessed with the 36-Item Short Form Health Survey (SF-36). The SF-36 evaluates 8 different domains of quality of life, i.e., physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The score of each domain ranges from 0 to 100, with high score indicating better function.

OTHER OUTCOMES:
Alterations of sleep architecture | During the night of surgery
  Sleep architecture is monitored with polysomnograph from 21:00 pm in the night of surgery to 06:00 am on the first day after surgery in part of enrolled patients (selected according to randomization block).
The Numeric Rating Scale (NRS) pain score within 5 days after surgery. | At 2, 6, 24, 48, 72, 96, and 120 hours (i.e., the 5th day) after surgery.
  The Numeric Rating Scale (NRS) pain score is assessed with the NRS (an 11-point scale where 0=no pain and 10=the worst pain).
Subjective sleep quality within 5 days after surgery | During the first 5 days after surgery
  Subjective sleep quality is assessed with NRS (an 11-point scale where 0=the best sleep and 10=the worst sleep) once daily (8:00-10:00 am) during postoperative days 1-5.
Daily prevalence of delirium during postoperative days 1-5 | During the first 5 days after surgery
  Daily prevalence of delirium during postoperative days 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Beijing University First Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crocker E, Beggs T, Hassan A, Denault A, Lamarche Y, Bagshaw S, Elmi-Sarabi M, Hiebert B, Macdonald K, Giles-Smith L, Tangri N, Arora RC. Long-Term Effects of Postoperative Delirium in Patients Undergoing Cardiac Operation: A Systematic Review. Ann Thorac Surg. 2016 Oct;102(4):1391-9. doi: 10.1016/j.athoracsur.2016.04.071. Epub 2016 Jun 22. PMID 27344279
- [Background] Gosselt AN, Slooter AJ, Boere PR, Zaal IJ. Risk factors for delirium after on-pump cardiac surgery: a systematic review. Crit Care. 2015 Sep 23;19(1):346. doi: 10.1186/s13054-015-1060-0. PMID 26395253
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Mu DL, Li LH, Wang DX, Li N, Shan GJ, Li J, Yu QJ, Shi CX. High postoperative serum cortisol level is associated with increased risk of cognitive dysfunction early after coronary artery bypass graft surgery: a prospective cohort study. PLoS One. 2013 Oct 15;8(10):e77637. doi: 10.1371/journal.pone.0077637. eCollection 2013. PMID 24143249
- [Background] Kamdar BB, Niessen T, Colantuoni E, King LM, Neufeld KJ, Bienvenu OJ, Rowden AM, Collop NA, Needham DM. Delirium transitions in the medical ICU: exploring the role of sleep quality and other factors. Crit Care Med. 2015 Jan;43(1):135-141. doi: 10.1097/CCM.0000000000000610. PMID 25230376
- [Background] Reade MC, Finfer S. Sedation and delirium in the intensive care unit. N Engl J Med. 2014 Jan 30;370(5):444-54. doi: 10.1056/NEJMra1208705. No abstract available. PMID 24476433
- [Background] Delaney LJ, Van Haren F, Lopez V. Sleeping on a problem: the impact of sleep disturbance on intensive care patients - a clinical review. Ann Intensive Care. 2015 Feb 26;5:3. doi: 10.1186/s13613-015-0043-2. eCollection 2015. PMID 25852963
- [Background] Korompeli A, Muurlink O, Kavrochorianou N, Katsoulas T, Fildissis G, Baltopoulos G. Circadian disruption of ICU patients: A review of pathways, expression, and interventions. J Crit Care. 2017 Apr;38:269-277. doi: 10.1016/j.jcrc.2016.12.006. Epub 2016 Dec 13. PMID 28012425
- [Background] Fanfulla F, Ceriana P, D'Artavilla Lupo N, Trentin R, Frigerio F, Nava S. Sleep disturbances in patients admitted to a step-down unit after ICU discharge: the role of mechanical ventilation. Sleep. 2011 Mar 1;34(3):355-62. doi: 10.1093/sleep/34.3.355. PMID 21358853
- [Background] Elliott R, McKinley S, Cistulli P, Fien M. Characterisation of sleep in intensive care using 24-hour polysomnography: an observational study. Crit Care. 2013 Mar 18;17(2):R46. doi: 10.1186/cc12565. PMID 23506782
- [Background] McPherson JA, Wagner CE, Boehm LM, Hall JD, Johnson DC, Miller LR, Burns KM, Thompson JL, Shintani AK, Ely EW, Pandharipande PP. Delirium in the cardiovascular ICU: exploring modifiable risk factors. Crit Care Med. 2013 Feb;41(2):405-13. doi: 10.1097/CCM.0b013e31826ab49b. PMID 23263581
- [Background] Leung JM, Sands LP, Newman S, Meckler G, Xie Y, Gay C, Lee K. Preoperative Sleep Disruption and Postoperative Delirium. J Clin Sleep Med. 2015 Aug 15;11(8):907-13. doi: 10.5664/jcsm.4944. PMID 25979094
- [Background] Roggenbach J, Klamann M, von Haken R, Bruckner T, Karck M, Hofer S. Sleep-disordered breathing is a risk factor for delirium after cardiac surgery: a prospective cohort study. Crit Care. 2014 Sep 5;18(5):477. doi: 10.1186/s13054-014-0477-1. PMID 25189637
- [Background] Papaioannou V, Mebazaa A, Plaud B, Legrand M. 'Chronomics' in ICU: circadian aspects of immune response and therapeutic perspectives in the critically ill. Intensive Care Med Exp. 2014 Dec;2(1):18. doi: 10.1186/2197-425X-2-18. Epub 2014 May 14. PMID 26266918
- [Background] Alamili M, Bendtzen K, Lykkesfeldt J, Rosenberg J, Gogenur I. Melatonin suppresses markers of inflammation and oxidative damage in a human daytime endotoxemia model. J Crit Care. 2014 Feb;29(1):184.e9-184.e13. doi: 10.1016/j.jcrc.2013.09.006. Epub 2013 Oct 17. PMID 24140166
- [Background] Keating GM. Dexmedetomidine: A Review of Its Use for Sedation in the Intensive Care Setting. Drugs. 2015 Jul;75(10):1119-30. doi: 10.1007/s40265-015-0419-5. PMID 26063213
- [Background] Mantz J, Josserand J, Hamada S. Dexmedetomidine: new insights. Eur J Anaesthesiol. 2011 Jan;28(1):3-6. doi: 10.1097/EJA.0b013e32833e266d. PMID 20881501
- [Background] Li Y, Wang B, Zhang LL, He SF, Hu XW, Wong GT, Zhang Y. Dexmedetomidine Combined with General Anesthesia Provides Similar Intraoperative Stress Response Reduction When Compared with a Combined General and Epidural Anesthetic Technique. Anesth Analg. 2016 Apr;122(4):1202-10. doi: 10.1213/ANE.0000000000001165. PMID 26991622
- [Background] Chen Z, Tang R, Zhang R, Jiang Y, Liu Y. Effects of dexmedetomidine administered for postoperative analgesia on sleep quality in patients undergoing abdominal hysterectomy. J Clin Anesth. 2017 Feb;36:118-122. doi: 10.1016/j.jclinane.2016.10.022. Epub 2016 Dec 1. PMID 28183547
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Wanat M, Fitousis K, Boston F, Masud F. Comparison of dexmedetomidine versus propofol for sedation in mechanically ventilated patients after cardiovascular surgery. Methodist Debakey Cardiovasc J. 2014 Apr-Jun;10(2):111-7. doi: 10.14797/mdcj-10-2-111. PMID 25114763
- [Background] Skrupky LP, Drewry AM, Wessman B, Field RR, Fagley RE, Varghese L, Lieu A, Olatunde J, Micek ST, Kollef MH, Boyle WA. Clinical effectiveness of a sedation protocol minimizing benzodiazepine infusions and favoring early dexmedetomidine: a before-after study. Crit Care. 2015 Apr 2;19(1):136. doi: 10.1186/s13054-015-0874-0. PMID 25887495
- [Background] Cruickshank M, Henderson L, MacLennan G, Fraser C, Campbell M, Blackwood B, Gordon A, Brazzelli M. Alpha-2 agonists for sedation of mechanically ventilated adults in intensive care units: a systematic review. Health Technol Assess. 2016 Mar;20(25):v-xx, 1-117. doi: 10.3310/hta20250. PMID 27035758
- [Background] Pasin L, Landoni G, Nardelli P, Belletti A, Di Prima AL, Taddeo D, Isella F, Zangrillo A. Dexmedetomidine reduces the risk of delirium, agitation and confusion in critically Ill patients: a meta-analysis of randomized controlled trials. J Cardiothorac Vasc Anesth. 2014 Dec;28(6):1459-66. doi: 10.1053/j.jvca.2014.03.010. Epub 2014 Jul 14. PMID 25034724
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Skrobik Y, Duprey MS, Hill NS, Devlin JW. Low-Dose Nocturnal Dexmedetomidine Prevents ICU Delirium. A Randomized, Placebo-controlled Trial. Am J Respir Crit Care Med. 2018 May 1;197(9):1147-1156. doi: 10.1164/rccm.201710-1995OC. PMID 29498534
- [Background] Eremenko AA, Chernova EV. [Dexmedetomidine use for intravenous sedation and delirium treatment during early postoperative period in cardio-surgical patients]. Anesteziol Reanimatol. 2013 Sep-Oct;(5):4-8. Russian. PMID 24624849
- [Background] Park JB, Bang SH, Chee HK, Kim JS, Lee SA, Shin JK. Efficacy and safety of dexmedetomidine for postoperative delirium in adult cardiac surgery on cardiopulmonary bypass. Korean J Thorac Cardiovasc Surg. 2014 Jun;47(3):249-54. doi: 10.5090/kjtcs.2014.47.3.249. Epub 2014 Jun 5. PMID 25207222
- [Background] Ji F, Li Z, Nguyen H, Young N, Shi P, Fleming N, Liu H. Perioperative dexmedetomidine improves outcomes of cardiac surgery. Circulation. 2013 Apr 16;127(15):1576-84. doi: 10.1161/CIRCULATIONAHA.112.000936. Epub 2013 Mar 19. PMID 23513068
- [Background] Li X, Yang J, Nie XL, Zhang Y, Li XY, Li LH, Wang DX, Ma D. Impact of dexmedetomidine on the incidence of delirium in elderly patients after cardiac surgery: A randomized controlled trial. PLoS One. 2017 Feb 9;12(2):e0170757. doi: 10.1371/journal.pone.0170757. eCollection 2017. PMID 28182690
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339